CLINICAL TRIAL: NCT06518733
Title: Orthodontic Treatment Impact on Day-to-Day Life Experience of Adolescents With Fixed Orthodontic Appliances: A Cross-Sectional Study
Brief Title: Orthodontic Treatment Impact on Life Experience of Adolescents With Fixed Orthodontic Appliances
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shimaa Mohamed Gaber, Master candidate, Cairo University
Other Study IDs: 11543267
Record Dates: First submitted 2024-07-17; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Orthodontic Appliance Complication

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Group A: patients with fixed labial orthodontic appliance
  Interventions: Other: appliance type
- Group B: patients with fixed labial appliance with palatal appliances
  Interventions: Other: appliance type
- Group C: patients with fixed labial appliance with miniscrews
  Interventions: Other: appliance type
- Group D: patients with fixed labial appliance with both palatal appliances and miniscrews
  Interventions: Other: appliance type
- Group E: patients with fixed retainer
  Interventions: Other: appliance type

INTERVENTIONS:
Other: appliance type — different types of appliances: labial fixed appliances only, fixed retainers, palatal appliances and miniscrews

SUMMARY:
This cross-sectional study aimed to investigate the impact of different fixed orthodontic appliances on the day-to-day life experience of adolescent patients at any stage of their orthodontic treatment. A validated questionnaire was translated and used in the assessment, 364 patients (242 female and 122 male) were recruited, impact on the social and emotional well-being status of the participants was assessed as well as oral health, pain, and discomfort.

DETAILED DESCRIPTION:
This cross-sectional study aimed to evaluate the impact of orthodontic treatment on the daily life experience of adolescents wearing fixed orthodontic appliances. We aimed to assess the impact of different fixed orthodontic appliances in a sample of 364 patients either having labial fixed orthodontic appliances only or combined with palatal anchorage appliances, combined with mini-screws, combined with both palatal anchorage appliances and mini-screws or having fixed retainers. The outcomes were the impact on the patient's social and emotional well-being status and the impact on the patient's oral health, pain, and discomfort. a questionnaire was distributed and the patient was asked to fill it in. The questionnaire is composed of 22 questions with a 3-point scale.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients
* Patients wearing fixed orthodontic appliances at any stage of treatment (labial fixed appliance only - labial fixed appliance combined with any palatal or lingual appliance - labial fixed appliance combined with mini-screws) or fixed retainers either in the upper arch only, lower arch only, or in both arches.
* Age: 13-18 years old

Exclusion Criteria:

* Patients who refused to participate in the study.
* Patients with cleft lip or palate.
* Illiterate patients.
* Patients who had a complicated medical history.
* Patients with severe skeletal discrepancy undergoing combined orthodontic and orthognathic surgical treatment.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Egyptian adolescent patients with age 13-18 with fixed orthodontic appliances
Sampling Method: Non-Probability Sample
Enrollment: 364 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Impact on the social and emotional well-being status of the patient. | during the intervention
  impact social and emotional well-being status of the patient is assessed using a questionnaire

SECONDARY OUTCOMES:
Impact on the oral health, pain, and discomfort of the respondent | during the intervention
  Impact on the oral health, pain, and discomfort of the respondent is assessed using a questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided